CLINICAL TRIAL: NCT04729270
Title: Treatment of Neck Pain With Transcranial Direct Current Stimulation: A Single Blind Randomized Controlled Trial
Brief Title: Treatment of Neck Pain With Transcranial Direct Current Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cadiz (Other)
Responsible Party: Principal Investigator, Manuel Rodriguez Huguet, Clinical professor, University of Cadiz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: tDCS
Record Dates: First submitted 2021-01-24; First posted 2021-01-28 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Cervical Syndrome
Keywords: Neck Pain; Physical Therapy Modalities; Manual Therapy; massage; Transcranial Direct Current Stimulation; Transcutaneous electrical nerve stimulation
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: RANDOMIZED CLINICAL TRIAL WITH BLIND EVALUATION BY THIRD PARTIES, LONGITUDINAL AND PROSPECTIVE.
Who Masked: Investigator
Masking Description: Blind researcher
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPERIMENTAL GROUP (Experimental): The intervention for this group consisted of 10 sessions with Transcranial Direct Current Stimulation for a month.
  Interventions: Procedure: Physiotherapy treatment with physium device.
- CONTROL GROUP (Experimental): The intervention for this group consisted of 10 sessions with Transcutaneous Electrical Nerve Stimulation (TENS) for a month.
  Interventions: Procedure: Conventional physiotherapy treatment.

INTERVENTIONS:
Procedure: Physiotherapy treatment with physium device. — The intervention for this group consisted of 10 sessions with Transcranial Direct Current Stimulation for a month.
  Arms: EXPERIMENTAL GROUP
Procedure: Conventional physiotherapy treatment. — The intervention for this group consisted of 10 sessions with Electrical Nerve Stimulation (TENS) for a month.
  Arms: CONTROL GROUP

SUMMARY:
This study aim to investigate the effects of Transcranial Direct Current Stimulation for improving pressure pain thresholds (PPTs), range of motion,Neck Disability Index, the multidimensional health related quality of life (SF-12) and the multidimensional health related quality of life and pain in patients with mechanical neck pain (NP).

DETAILED DESCRIPTION:
Fifty-four participants with NP will randomly allocated to either an Transcranial Direct Current Stimulation (ten sessions) or transcutaneous electric nerve stimulation (TENS) (ten sessions) during two weeks. . Visual Analogue Scale (VAS), Neck Disability Index ( NDI), range of motion and (CROM), Questionnaire SF-12 and PPTs in sub-occipital and upper trapezius muscles were measured at baseline, at the end of treatment and at 1 month follow-up. T-tests and a repeated-measures multivariate analysis of variance (RM-MANOVA) were used for VAS, CROM and PPTs, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes,
* Aged between 18 and 60 years, in an
* Active state of pain and diagnosed with a month of evolution.

Exclusion Criteria:

- Patients who are pregnant, have pacemaker and those Surgically operated cervical spine - Patients who have been treated with Transcranial Direct Current Stimulation a month earlier.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
The intensity of cervical pain | Baseline
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patients' current level of cervical pain, and the worst and lowest level of pain experienced in the preceding week in the cervical area.

SECONDARY OUTCOMES:
The intensity of cervical pain | Four weeks
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patients' current level of cervical pain, and the worst and lowest level of pain experienced in the preceding week in the cervical area.
The intensity of cervical pain | Twelve weeks
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patients' current level of cervical pain, and the worst and lowest level of pain experienced in the preceding week in the cervical area.
Active cervical range of motion | Baseline,four weeks and Twelve weeks.
  Measured by goniometer type crom
Pressure pain thresholds in cervical trigger points | Baseline,four weeks and Twelve weeks.
  Pressure pain thresholds (PPTs) will be measured with a pressure algometer (Baseline,
Neck Disability Index (NDI). | Baseline,four weeks and Twelve weeks.
  Questionnaire Neck Disability Index (NDI).

CONTACTS AND LOCATIONS:
Overall Officials: manuel Rodríguez Huguet, Physiotherapy, Principal Investigator — University of Cádiz
Locations (1):
- Policlínica Santa María, Cadiz, Cádiz, Spain

REFERENCES:
- [Background] Whiteford CM, Steinbeck L, Dommerholt J. On "Clinical Practice Guideline for Physical Therapy Assessment and Treatment in Patients With Nonspecific Neck Pain," Bier JD, Scholten-Peeters WGM, Staal JB, et al. Phys Ther. 2018;98:162-171. Phys Ther. 2018 Sep 1;98(9):819-820. doi: 10.1093/ptj/pzy078. No abstract available. PMID 29961845
- [Background] Cohen SP. Epidemiology, diagnosis, and treatment of neck pain. Mayo Clin Proc. 2015 Feb;90(2):284-99. doi: 10.1016/j.mayocp.2014.09.008. PMID 25659245
- [Background] Cohen SP, Hooten WM. Advances in the diagnosis and management of neck pain. BMJ. 2017 Aug 14;358:j3221. doi: 10.1136/bmj.j3221. PMID 28807894
- [Background] Blanpied PR, Gross AR, Elliott JM, Devaney LL, Clewley D, Walton DM, Sparks C, Robertson EK. Neck Pain: Revision 2017. J Orthop Sports Phys Ther. 2017 Jul;47(7):A1-A83. doi: 10.2519/jospt.2017.0302. PMID 28666405
- [Background] Cote P, Yu H, Shearer HM, Randhawa K, Wong JJ, Mior S, Ameis A, Carroll LJ, Nordin M, Varatharajan S, Sutton D, Southerst D, Jacobs C, Stupar M, Taylor-Vaisey A, Gross DP, Brison RJ, Paulden M, Ammendolia C, Cassidy JD, Loisel P, Marshall S, Bohay RN, Stapleton J, Lacerte M. Non-pharmacological management of persistent headaches associated with neck pain: A clinical practice guideline from the Ontario protocol for traffic injury management (OPTIMa) collaboration. Eur J Pain. 2019 Jul;23(6):1051-1070. doi: 10.1002/ejp.1374. Epub 2019 Feb 28. PMID 30707486
- [Background] Fitzgibbon BM, Schabrun SM. Transcranial Direct Current Stimulation for Pain Disorders: Challenges and New Frontiers. Clin Pharmacol Ther. 2019 Oct;106(4):717-719. doi: 10.1002/cpt.1544. Epub 2019 Jul 15. No abstract available. PMID 31309544
- [Background] Yalinay Dikmen P, Yavuz BG, Aydinlar EI. The relationships between migraine, depression, anxiety, stress, and sleep disturbances. Acta Neurol Belg. 2015 Jun;115(2):117-22. doi: 10.1007/s13760-014-0312-0. Epub 2014 Jun 3. PMID 24889393
- [Background] Schwartz DP, Robbins MS. Primary headache disorders and neuro-ophthalmologic manifestations. Eye Brain. 2012 Sep 13;4:49-61. doi: 10.2147/EB.S21841. eCollection 2012. PMID 28539781
- [Background] Nitsche MA, Paulus W. Transcranial direct current stimulation--update 2011. Restor Neurol Neurosci. 2011;29(6):463-92. doi: 10.3233/RNN-2011-0618. PMID 22085959
- [Background] Martelletti P, Jensen RH, Antal A, Arcioni R, Brighina F, de Tommaso M, Franzini A, Fontaine D, Heiland M, Jurgens TP, Leone M, Magis D, Paemeleire K, Palmisani S, Paulus W, May A; European Headache Federation. Neuromodulation of chronic headaches: position statement from the European Headache Federation. J Headache Pain. 2013 Oct 21;14(1):86. doi: 10.1186/1129-2377-14-86. PMID 24144382
- [Background] Charvet LE, Shaw MT, Bikson M, Woods AJ, Knotkova H. Supervised transcranial direct current stimulation (tDCS) at home: A guide for clinical research and practice. Brain Stimul. 2020 May-Jun;13(3):686-693. doi: 10.1016/j.brs.2020.02.011. Epub 2020 Feb 10. PMID 32289698
- [Background] Caulfield KA, Badran BW, DeVries WH, Summers PM, Kofmehl E, Li X, Borckardt JJ, Bikson M, George MS. Transcranial electrical stimulation motor threshold can estimate individualized tDCS dosage from reverse-calculation electric-field modeling. Brain Stimul. 2020 Jul-Aug;13(4):961-969. doi: 10.1016/j.brs.2020.04.007. Epub 2020 Apr 21. PMID 32330607
- [Background] DaSilva AF, Truong DQ, DosSantos MF, Toback RL, Datta A, Bikson M. State-of-art neuroanatomical target analysis of high-definition and conventional tDCS montages used for migraine and pain control. Front Neuroanat. 2015 Jul 15;9:89. doi: 10.3389/fnana.2015.00089. eCollection 2015. PMID 26236199
- [Background] Auvichayapat P, Janyacharoen T, Rotenberg A, Tiamkao S, Krisanaprakornkit T, Sinawat S, Punjaruk W, Thinkhamrop B, Auvichayapat N. Migraine prophylaxis by anodal transcranial direct current stimulation, a randomized, placebo-controlled trial. J Med Assoc Thai. 2012 Aug;95(8):1003-12. PMID 23061303
- [Background] Straudi S, Buja S, Baroni A, Pavarelli C, Pranovi G, Fregni F, Basaglia N. The effects of transcranial direct current stimulation (tDCS) combined with group exercise treatment in subjects with chronic low back pain: a pilot randomized control trial. Clin Rehabil. 2018 Oct;32(10):1348-1356. doi: 10.1177/0269215518777881. Epub 2018 May 21. PMID 29783893
- [Background] Andrade SM, de Brito Aranha REL, de Oliveira EA, de Mendonca CTPL, Martins WKN, Alves NT, Fernandez-Calvo B. Transcranial direct current stimulation over the primary motor vs prefrontal cortex in refractory chronic migraine: A pilot randomized controlled trial. J Neurol Sci. 2017 Jul 15;378:225-232. doi: 10.1016/j.jns.2017.05.007. Epub 2017 May 3. PMID 28566169
- [Background] Przeklasa-Muszynska A, Kocot-Kepska M, Dobrogowski J, Wiatr M, Mika J. Transcranial direct current stimulation (tDCS) and its influence on analgesics effectiveness in patients suffering from migraine headache. Pharmacol Rep. 2017 Aug;69(4):714-721. doi: 10.1016/j.pharep.2017.02.019. Epub 2017 Mar 1. PMID 28551531